CLINICAL TRIAL: NCT04316702
Title: Hyperbaric Oxygen Therapy vs. Pharmaceutical Therapy in Patients Suffering From Fibromyalgia That Was Induced by Emotional Trauma: Prospective, Randomized, Two Active Arms Clinical Trial
Brief Title: Hyperbaric Oxygen Therapy Compared to Pharmaceutical in Fibromyalgia With Emotional Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: The Emili Sagol Creative Arts Therapies Research Center (Unknown)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Head of Sagol center for hyperbaric medicine and research, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ASF-20-0008
Record Dates: First submitted 2020-03-03; First posted 2020-03-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia; Emotional Trauma
MeSH Terms: conditions — Fibromyalgia | interventions — Hyperbaric Oxygenation; Therapeutics; Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: randomized controlled trial using conventional pharmacotherapy treatment compared to hyperbaric oxygen therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: randomization by computer, the patient and her primary care physician will know the treatment received. Any side effects during therapy will be reported to the care providers and nurses and physicians unrelated to the study. Investigators and outcome assessors will not know the patient's arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Oxygen (Active Comparator): 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week. Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Interventions: Device: Hyperbaric oxygen therapy (HBOT) treatment
- Pharmacotherapy (Active Comparator): Two medications currently licensed for the treatment of FM in Israel, i.e. Cymbalta and Lyrica. Treatment with Lyrica will start at a dose of 75 mg twice a day, at morning and at bedtime, while treatment with Cymbalta will start at a dose of 30 mg a day (in the morning). After a period of 2 weeks, patients will be evaluated and dose will be adjusted as necessary and tolerated, up to the maximum dosage recommended for FM. Patients may also be switched from one medication to the other according to clinical judgment of the physician.
  Interventions: Drug: Cymbalta / Lyrica - Drug treatment

INTERVENTIONS:
Device: Hyperbaric oxygen therapy (HBOT) treatment — 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week. Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Arms: Hyperbaric Oxygen
Drug: Cymbalta / Lyrica - Drug treatment — one of the two medications currently licensed for the treatment of FMS in Israel, i.e. Cymbalta and Lyrica. Two medications currently licensed for the treatment of FM in Israel, i.e. Cymbalta and Lyrica. Treatment with Lyrica will start at a dose of 75 mg twice a day, at morning and at bedtime, while treatment with Cymbalta will start at a dose of 30 mg a day (in the morning).
  Arms: Pharmacotherapy

SUMMARY:
The investigators have previously studied the efficacy of hyperbaric oxygen therapy (HBOT) as a treatment for Fibromyalgia syndrome (FMS) in a prospective, active control, crossover clinical trial. The results demonstrated significant amelioration of all FMS symptoms, with significant improvement in life quality; furthermore, the investigators were able to demonstrate significant neuroplasticity on SPECT imaging, with a decrease of the hyperactivity in posterior regions and elevation of the reduced activity in frontal areas.

In this study, the investigators intend to both repeat and expand the investigator's previous findings, treating FMS patients with history of emotional trauma with HBOT, while performing an extensive of evaluation both before and after treatment.

In the current study, the investigators plan to compare HBOT to current standard of care of FMS (pharmacological and non - pharmacological).

DETAILED DESCRIPTION:
The study will include 60 fibromyalgia patients in whom emotional trauma, such as childhood abuse, could be considered as the trigger for FMS. Each participant will be examined at the time of recruitment and a diagnosis of FMS will be verified, based on the updated 2016 diagnostic criteria. In the current study the investigators will recruit patients not currently being treated with the target medications (Lyrica or Cymbalta).

Patients will undergo randomization upon recruitment to one of the two study groups. One group will proceed to a course of HBOT treatment while the second group will commence with standard treatment for FMS, as outlined in the Israeli guidelines for the diagnosis and treatment of FMS .

HBOT protocol: a total of 60 daily hyperbaric oxygen treatment sessions will be administrated 5 days per week. 60 sessions will include exposure of 90 minutes to 100% at 2 Absolute atmospheres (ATA), with 5 minutes air breaks every 20 minutes.

Pharmaceutical protocol: patients will be offered pharmacological treatment with one of the two medications currently licensed for the treatment of FMS in Israel, i.e. Cymbalta and Lyrica. Treatment with Lyrica will start at a dose of 75 mg twice a day, at morning and at bedtime, while treatment with Cymbalta will start at a dose of 30 mg a day (in the morning). After a period of 2 weeks, patients will be evaluated and dose will be adjusted as necessary and tolerated, up to the maximum dosage recommended for FM. Patients may also be switched from one medication to the other according to clinical judgment of the physician.

ELIGIBILITY:
Inclusion Criteria:

* FM diagnosis based on the widespread pain index (WPI) and the Symptom Severity Score (SSS).
* Score at the trauma questionnaire indicating low, moderate or severe trauma in one of the criteria specified in the questionnaire.
* Ability to provide informed consent
* Age>18

Exclusion Criteria:

* Presence of systemic inflammatory disorders including inflammatory rheumatological and autoimmune disorders.
* History of traumatic brain injury (TBI)
* Other FM etiologies
* Currently or previously treated with Duloxetine (Cymbalta) or Pregabalin (Lyrica)
* Contraindications to both Lyrica and Cymbalta
* Major psychiatric disorder (such as major depression, schizophrenia, bi-polar disorder)
* Previous suicidal attempt/s
* Does not take part in psychotherapy on a weekly basis (minimum)
* Previous HBOT for any other reason prior to their inclusion
* Chest pathology (including active asthma)
* Inner ear disease
* Claustrophobia
* Inability to perform awake brain MRI test
* Chronic renal failure (eGFR< 60 ml/min)
* Previous neurological conditions (eg. Epilepsy, neuromuscular diseases, metabolic diseases, etc.); Brain tumors; Skull base fractures; Active malignancy; s/p neurosurgery
* Active Smoking
* Pregnancy or not committing to not getting pregnant during the study period

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) questionnaire | at 3 months
  Fibromyalgia Impact Questionnaire (FIQ) questionnaire score at the end of treatment period (HBOT/pharmaceutical). Score range 0-100, higher score means worse outcome
Fibromyalgia Impact Questionnaire (FIQ) questionnaire | at 6 months
  Fibromyalgia Impact Questionnaire (FIQ) questionnaire score at the end of follow up period (HBOT/pharmaceutical). Score range 0-100, higher score means worse outcome

SECONDARY OUTCOMES:
Widespread pain index questionnaire | at baseline, 3 months, 6 months
  Fibromyalgia syndrome symptoms questionnaire named:Wide Spread Pain Index (scale 0-19, higher score means worse outcome)
Symptoms severity scale questionnaire | at baseline, 3 months, 6 months
  Fibromyalgia syndrome symptoms questionnaire named:Symptom Severity Scale (SSS) (scale 0-12, higher score means worse outcome)
Post traumatic stress disorder (PTSD) symptoms scale (PSS) questionnaire | at baseline, 3 months, 6 months
  a 17-item semi-structured interview that assesses the presence and severity of Diagnostic and Statistical Manual (DSM-IV) PTSD symptoms related to a single identified traumatic event in individuals with a known trauma history. scale 0-51, higher score means worse outcome
Medical somatic dissociation questionnaire (MSDQ) | at baseline, 3 months, 6 months
  assess somatic dissociation in the healthcare system setting, Scale 5-130, higher score means worse outcome
Recovery promoting relationships scale (RPRS) | at baseline, 3 months, 6 months
  assesses patient-therapist relationships from the patient's perspective.
the brief symptom inventory (BSI-18) | at baseline, 3 months, 6 months
  evaluate psychological distress, three sub-scales: depression, anxiety, and somatization. scale of 0-24, higher score means worse outcome.
Beck depression inventory (BDI) | at baseline, 3 months, 6 months
  a 21-question multiple choice self-report inventory, designed to measure severity of depression. scale of 0-63, higher score means worse outcome
Short form health survey (sf-36) | at baseline, 3 months, 6 months
  Quality of life questionnaire, scale of 0-100, higher score means better outcome
patient's global impression of change PGIC questionnaire | at 3 months, at 6 months
  patient's global impression of change questionnaire, scale of 1-7, higher score means better outcome
draw a person (DAP) assignment | at baseline, 3 months, 6 months
  self drawing tool, allows the expression of hidden or repressed thoughts and feelings in a relatively rapid and simple way by passing the censorship defensive mechanism
Heat pain threshold | at baseline, 3 months
  Heat pain threshold is determined as the minimum temperature causing pain. Thermal pain is induced with thermal electrode (thermode). Thermode temperature will initially be set at 32.0°C and gradually increase at a rate of 0.3°C/sec. Participants will be instructed to report when the sensation produced by the thermode changed from heat sensation to pain (heat-pain threshold). This procedure will be conducted three times for every subject and the mean of the trials will be calculated.
conditioned pain modulation using Heat test-stimulus (HTS) | at baseline, 3 months
  Following heat pain thresholds assessments, the thermode will be applied on the forearm for 120 seconds at constant temperature. The temperature will be individually adapted to induce a mean pain intensity of 50/100, Participant's pain intensity will be evaluated by numeric pain rating scale (NPRS) ranging from 0 (no pain) to 100 (most intense pain tolerable). The 120-second HTS will be done before and during cold water immersion of the contralateral hand in 10 Celsius degrees, using the same thermode temperature to measure conditioned pain modulation (CPM). CPM efficiency will be evaluated by computing the difference in mean pain intensity induced by the pressure stimulus and the Heat test-stimulus (HTS) before and during the Cold water immersion of the opposite hand. Thus, effective pain inhibitory mechanisms are represented by higher (positive) values
Cerebral blood volume | at baseline, 3 months
  Cerebral blood volume (in milliliter) will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
Cerebral blood Flow | at baseline, 3 months
  Cerebral blood volume (in milliliter/min) will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
Fractional anisotropy | at baseline, 3 months
  Brain microstructure imaging will evaluate fractional anisotropy (FA , scale 0-1 in each region of interest. The MRI protocol will include diffusion tensor imaging (DTI)
Mean diffusivity | at baseline, 3 months
  Brain microstructure imaging will evaluate mean diffusivity (MD, scale 0-1 in each region of interest. The MRI protocol will include diffusion tensor imaging (DTI).
Brain function imaging | at baseline, 3 months
  Resting state fMRI(rsfMRI or R-fMRI)- a method of functional brain imaging that can be used to evaluate regional interactions that occur when a subject is not performing an explicit task. This resting brain activity is observed through changes in blood flow in the brain which creates what is referred to as a blood-oxygen-level dependent (BOLD) signal that can be measured using functional Magnetic Resonance Imaging (fMRI).
Metabolic Brain function imaging | at baseline, 3 months
  Brain Single photon emission computed tomography (SPECT) will be conducted.
Brain functionality | at baseline, 3 months
  FMRI tasks will evaluate brain function during cognitive (working memory task) and emotional tasks (emotion recognition task)
NeuroTrax | at baseline, 3 months
  computerized cognitive evaluation battery
CANTAB Cambridge Neuropsychological Test Automated Battery | at baseline, 3 months
  computerized cognitive evaluation battery
Physical activity | at baseline, 3 months
  The daily physical activity will be objectively tracked by Garmin watch technology. The watch will be also wired during night for measurements of the time asleep, restless and awake, trackers help you understand each night to make the most of each day
Inflammatory cytokines | at baseline, 3 months
  Blood Tests will include: IL-1, IL-6, Tumor necrosis factor-alpha, C-reactive protein (CRP).
Endocrine system | at baseline, 3 months
  Free cortisol, Adrenocorticotropic hormone (ACTH) in blood tests and a hair sample for cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- hyperbaric center Asaf harofe medical center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: No